CLINICAL TRIAL: NCT04905940
Title: Evaluation of Cost-Effectiveness And Clinical Effectiveness of Mouthwash Containing Curcuma Longa Versus Essential Oil and A Placebo Mouthwash on Controlling Halitosis Among Egyptian Children: A Randomized Clinical Trial
Brief Title: Evaluation of Clinical and Cost-effectiveness of Different Mouthwashes on Controlling Halitosis Among a Group of Egyptian Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Mohammed Elsaeed Ahmed, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422019461401
Record Dates: First submitted 2021-05-19; First posted 2021-05-28 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Halitosis
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Turmeric mouthwash (Experimental): Evaluation of cost-effectiveness of turmeric mouthwash in controlling halitosis
  Interventions: Drug: Turmeric mouthwash
- Essential oil mouthwash (Active Comparator): Evaluation of cost-effectiveness of essential oil mouthwash in controlling halitosis
  Interventions: Drug: Turmeric mouthwash
- Placebo mouthwash (Placebo Comparator): Evaluation of cost-effectiveness of placebo mouthwash in controlling halitosis
  Interventions: Drug: Turmeric mouthwash

INTERVENTIONS:
Drug: Turmeric mouthwash — Turmeric mouthwash evaluation in controlling halitosis

SUMMARY:
To evaluate the clinical and cost-effectiveness of mouthwash containing Curcuma longa (Turmeric extract) versus mouthwash containing essential oils and Placebo mouthwash on controlling Halitosis among a group of Egyptian children.

DETAILED DESCRIPTION:
For both interventions:

1. Eligibility screen and patient selection according to the inclusion and exclusion criteria.
2. Readings for halitosis will be recorded using Tanita HC-312F Fitscan Portable Breath Checker (Tanita Corporation, Japan) that shows red, yellow and green colors indicating halitosis degree.

   * Green color=no odour
   * Yellow color=moderate odour
   * Red color=intense odour Children with yellow or red colored results will be included.
3. Participants will be provided with information regarding the risks and benefit of the study and written informed consent will be obtained.
4. Intra and extra-oral examinations and Baseline records photographs, caries assessment by using DMF, gingival condition assessment using Simplified oral hygiene index and personal data collection.
5. Participating children will be offered a full mouth restorative treatment, if needed, before starting the trial to exclude that halitosis comes from food impaction in carious teeth.
6. In another visit, after the full mouth rehabilitation, readings for halitosis will be re-recorded using color coded Tanita HC-312F Fitscan Portable Breath Checker (Tanita corporate, Japan). Patients who will get green colored result will be excluded from the study as the cause of halitosis in those patients would be food impaction in carious teeth.
7. Allocation of the participants who will score more than 2 into either one of three groups; A, B or C. i. A for Experimental group (Turmeric mouthwash) ii. B for first comparator (Essential oil mouthwash) iii. C for second comparator (Placebo)

   Allocation will be concealed by withdrawing a sealed opaque envelope containing four times folded paper containing the type of mouth wash that will be used. This will decrease performance bias as the operator will not know the group of the participant until taking the score of the patients and finishing the restorative treatment. Blinding of the operator will not be needed as the readings will be objective and recorded using the device (Tanita device) not by the operator (organoleptic method).
8. All mouth rinse samples (experimental and comparators 1&2) will be put into identical white opaque plastic bottles labelled with the codes A, B or C for the blinding of the participant. Group A: The experimental sample is a Turmeric mouthwash which will be prepared by dissolving 10 mg of Turmeric extract in 100 mL of distilled water and 0.005% of flavouring agent peppermint oil (Sharma, 2016). Group B: The first comparator will be the commercial Miswak Listerine mouthwash. Group C: The second comparator will be a placebo mouthwash and will be prepared with peppermint oil and distilled water; essentially the same contents as those in the experimental mouthwash except for the turmeric powder.
9. Every participant will use 2 mouthwash bottles of the same group label that they were allocated to. The first bottle according to their allocation. Patients will be given standard written oral hygiene instructions and mouth washing instructions to rinse twice daily with 10 ml for 1 minute under their parents" supervision for two weeks.
10. The first follow up visit after two weeks, the halitosis score will be recorded by using the Tanita device for numerical record and by asking the parent if there is a bad odour or not. Patients then will be instructed to stop rinsing for the next two weeks while maintaining other oral hygiene instructions.
11. The second follow-up visit after 4 weeks, patients will be given the second bottle and instructed to rinse twice daily with 10 ml for another two weeks.
12. The last follow up visit will be after 6 weeks and the final Halitosis score will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-12 years old.
* Cooperative children.
* Both genders.
* Medically free to exclude systemic cause of halitosis.
* Bad breath

Exclusion Criteria:

* Children using any other oral hygiene aid other than routine teeth brushing.
* Children with a known history of allergy to any mouthwash or drug.
* Parents refuse to participate in the trial.
* Treatment by antibiotic within one month before the trial(Pham & Nguyen, 2018).
* Abscess, draining sinus, cellulitis, or other conditions requiring emergency dental treatment.
* Children using fixed or removable orthodontic appliances or dentures.
* Children with a history of deleterious oral habits of mouth breathing.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Questionnaire for Patient related side effects | 45 days
  the measuring unit will be binary (yes/no) from the parent and child.
  While using the mouthwash:
  1. Is the Child's quality of life changed for the better?
  2. Acceptance and safety of the mouth wash

SECONDARY OUTCOMES:
Cost-effectiveness | 45 days
  Economic and Clinical effectiveness of turmeric mouthwash
  Cost effectiveness will be measured according to ICER (Incremental cost-effectiveness ratio)

IPD SHARING:
Plan to Share IPD: No